CLINICAL TRIAL: NCT06503692
Title: A Multicentre, Randomized Controlled Clinical Trial of Scoring Balloon Versus High Pressure Balloon in the Treatment of Arteriovenous Graft Stenosis
Brief Title: Scoring Balloon and High Pressure Balloon in the Treatment of Arteriovenous Graft Stenosis
Acronym: DKTAVG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DK Medical Technology (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR-0171
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Arteriovenous Graft Stenosis
Keywords: Arteriovenous Graft Stenosis; Scoring Balloon; Angioplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DKutting PTA Scoring Balloon Dilatation Catheter (Experimental): Subjects in this group are treated with DKutting PTA Scoring Balloon Dilatation Catheter
  Interventions: Device: DKutting PTA Scoring Balloon Dilatation Catheter
- Peripheral Balloon Catheter (Active Comparator): Subjects in this group are treated with Peripheral Balloon Catheter
  Interventions: Device: Peripheral Balloon Catheter

INTERVENTIONS:
Device: DKutting PTA Scoring Balloon Dilatation Catheter — The device consists of a balloon catheter with scoring elements (triangular cross-section) fixed to the surface of the balloon and distributed radially at every 120°. When the balloon is inflated, the expansion force is focused along the scoring elements, causing it to expand under lower balloon pressure.
  Other Names: Scoring Balloon
  Arms: DKutting PTA Scoring Balloon Dilatation Catheter
Device: Peripheral Balloon Catheter — The device is an over-the-wire (OTW) double-lumen balloon catheter. The balloon is inflated to a known diameter at a specified pressure.
  Arms: Peripheral Balloon Catheter

SUMMARY:
This is a multicenter, prospective, randomized controlled clinical study. Patients with hemodialysis arteriovenous graft fistula stenosis will be recruited to explore whether the scoring balloon is superior to the high pressure balloon in treating such lesions, so as to provide a basis for optimizing the treatment of such lesions.

This study will be conducted in seven (7) clinical trial institutions, with a total of 140 subjects included. After randomization, the subjects will use either the scoring balloon dilatation catheter, developed and produced by DK Medical Technology Co., Ltd., or the peripheral balloon dilatation catheter for surgical treatment. Clinical follow-up will be carried out within 5 days, 3 months, 6 months, and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodialysis patients aged ≥18 and ≤80 years old, (Note: Hemodialysis patients in Singapore aged ≥ 21 and ≤80 years old);
2. AVG is mature and has successfully completed at least one hemodialysis treatment;
3. The target lesion is located in the AVG return vein and the venous side anastomosis;
4. The degree of stenosis of the target lesion is ≥50% (DSA visual inspection), and one of the following clinical indicators exists at the same time: Physical examination abnormalities include: open collateral veins, ipsilateral limb edema, changes in pulse characteristics, abnormal tremors, abnormal murmurs, etc.; Dialysis abnormalities include: increased venous pressure, new puncture difficulties, aspiration of thrombi, inability to reach target dialysis blood flow, prolonged haemostasis time after needle removal for 3 consecutive times, unexplained decrease in dialysis dose Kt/V (>0.2 units), decrease in brachial artery blood flow (brachial artery blood flow <650ml/min or decreased by 20% compared with the previous follow-up visit), etc.
5. The target lesion is primary or restenotic, consisting of one or more series of lesions, and the reference blood vessel diameter of the target lesion is between 4.0-8.0mm, and the total length of the target lesion is ≤80mm ;
6. The patient voluntarily signs the informed consent form.

Exclusion Criteria:

1. The target lesion is located in the feeding artery, arterial anastomosis, artificial blood vessel puncture site, cephalic venous arch, thoracic outlet or central vein;
2. A stent has been implanted in any part of the access or there is ipsilateral central vein stenosis or occlusion that affects the function of the access;
3. Severely calcified lesions that are not expected to be dilatable with balloons;
4. Acute thrombosis or chronic total occlusion of AVG occurred at the time of enrolment;
5. The target lesion or any part of the vascular access has received PTA treatment within the last month;
6. There are thicker branch veins in the vein opening of the end-to-side anastomosis;
7. Patients who have undergone major surgical treatment within 30 days before inclusion in the study;
8. Patients known to be allergic to or intolerant to contrast media;
9. Patients receiving glucocorticoids or immunosuppressants;
10. The patient's life expectancy is less than 1 year;
11. Patients planning kidney transplantation or switching to peritoneal dialysis;
12. The degree of stenosis in the puncture point area is >50%；
13. Patients with infection or other medical conditions that make the investigator think they are not suitable to participate in this study;
14. Those who have participated in clinical trials of other drugs or devices but have not completed them.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Primary Patency (TLPP) at 6 months post-procedure | 6 months
  TLPP is terminated by postoperative target lesion failure (TLF) (including the 5 mm range before and after the target lesion) or target lesion-related vascular access thrombosis.
  TLF is defined as the presence of at least one clinical indicator (defined according to the NKF-K/DOQI guidelines) caused by target lesion stenosis ( ≥50% stenosis of the target lesion assessed by contrast angiography or ultrasound), including physical examination abnormalities or dialysis abnormalities.
  Target lesion-related vascular access thrombosis is limited to: after the thrombus is removed during AVG thrombus treatment and before balloon dilatation, it is confirmed by ultrasound/DSA that the original target lesion has a stenosis ≥ 50%, or when the balloon is expanded with low pressure (<6 atm) during intraluminal treatment, obvious balloon residual waisting can be seen at the target lesion; simple mural thrombus at the puncture point or other parts of the graft needs to be ruled out.

SECONDARY OUTCOMES:
Target Lesion Primary Patency (TLPP) at 12 months post-procedure | 12 months
  TLPP is terminated by postoperative target lesion failure (TLF) (including the 5 mm range before and after the target lesion) or target lesion-related vascular access thrombosis.
  TLF is defined as the presence of at least one clinical indicator (defined according to the NKF-K/DOQI guidelines) caused by target lesion stenosis ( ≥50% stenosis of the target lesion assessed by contrast angiography or ultrasound), including physical examination abnormalities or dialysis abnormalities.
  Target lesion-related vascular access thrombosis is limited to: after the thrombus is removed during AVG thrombus treatment and before balloon dilatation, it is confirmed by ultrasound/DSA that the original target lesion has a stenosis ≥ 50%, or when the balloon is expanded with low pressure (<6 atm) during intraluminal treatment, obvious balloon residual waisting can be seen at the target lesion; simple mural thrombus at the puncture point or other parts of the graft needs to be ruled out.
Access Circuit Primary Patency (ACPP) at 6 and 12 months post-procedure | 6, 12 months post-procedure
  ACPP is terminated when stenosis or thrombus causing abnormal clinical indicators occurs in any part of the AVG after surgery (inflow artery, entire graft, and outflow vein, including central vein). (Definition according to NKF- K/DOQI guidelines), including physical examination abnormalities or dialysis abnormalities. Physical examination abnormalities include: open collateral veins, ipsilateral limb edema, changes in pulse characteristics, abnormal tremors, abnormal murmurs, etc.; Dialysis abnormalities include: increased venous pressure, new puncture difficulties, aspiration of thrombi, inability to reach target dialysis blood flow, prolonged haemostasis time after needle removal for 3 consecutive times, unexplained decrease in dialysis dose Kt/V (>0.2 units), decrease in brachial artery blood flow (brachial artery blood flow <650ml/min or decreased by 20% compared with the previous follow-up visit), etc.
Access Circuit Secondary Patency (ACSP) 6 and 12 months after surgery | 6, 12 months post-procedure
  ACSP terminates when the AVG is abandoned due to various reasons after surgery, during which multiple interventions can be performed to maintain the patency of the entire pathway.
Acute Lumen Gain | During the procedure
  Immediately after dilation, DSA uses two different angles (≥45°) for angiography (a unified x-ray ruler will be provided as the reference object to reduce measurement errors) Calculation formula: minimum lumen diameter of the target lesion immediately after dilation - minimum lumen diameter of the target lesion before procedure.
Technical Success | 0-5 days post-procedure
  Residual stenosis of the target lesion after surgery is ≤30%, and no serious adverse events related to the investigational device occurred during the perioperative period.
Clinical Success | 0-5 days post-procedure
  Complete at least one successful hemodialysis session after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pei Wang, MD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (7):
- China (6):
  - Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - South China Hospital of Shenzhen University, Shenzhen, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
- National University Hospital of Singapore, Singapore, Singapore